CLINICAL TRIAL: NCT06442553
Title: New Generation Low Level Laser Effect on Masseter Muscle Oxygenation, Bite Force and Algometric Changes in Myofacial Pain Syndrome: A Randomised, Placebo-controlled Clinical Trial
Brief Title: New Generation Low Level Laser Effect in Myofacial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, İREM KARAGOZOGLU, Assist. Prof., University of Gaziantep
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: KARAGOZOGLUI
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Myofascial Pain Syndrome
Keywords: low level laser therapy; myofascial pain syndrome; bite forces; visual analogue scale; gaalas laser; neodymium doped yttrium aluminum garnet lasers
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GRR laser (Experimental): patients received 15 sessions GRR laser treatment for 3 weeks
  Interventions: Device: GRR laser
- Nd:YAG Laser (Experimental): patients received 10 sessions Nd:YAG laser treatment for 2 weeks
  Interventions: Device: Nd:YAG laser
- placebo (Placebo Comparator): patients received 10 sessions emission-free laser treatment for 2 weeks
  Interventions: Device: Nd:YAG laser

INTERVENTIONS:
Device: GRR laser — A total of 15 sessions were applied to each patient for three weeks, five times per week.
  Arms: GRR laser
Device: Nd:YAG laser — A total of 10 sessions, five sessions per week, were applied
  Arms: Nd:YAG Laser; placebo

SUMMARY:
Low level laser treatments have been used to treat painful trigger points in myofascial pain syndrome (MPS), but the effectiveness of the appropriate laser type and parameters is still uncertain. The aim of this study was to compare the effectiveness of different types of low level laser treatment (LLLT) in reducing pain levels, changing oxygen saturation and bite force in patients with MPS.

DETAILED DESCRIPTION:
A total of 45 patients with MPS were randomly divided into three groups. First group received LLLT with GRR laser over massater muscle region. Patients in the second group were treated with Nd:YAG laser and the same protocol with Nd:YAG laser was performed in the placebo group using sham device. Pain was evaluated by visual analogue scale (VAS), change in oxygen concentration in the massater muscle was measured by functional near-infrared spectroscopy- fNIRS and bite force was measured with Flexiforce sensors before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

-patients with symptoms of temporomandibular disorders and diagnosed with MPS as a result of the clinical examination.

Exclusion Criteria:

* Patients with internal TMJ irregularities or degenerative joint changes,
* patients with restricted mouth opening, deviation or deflection,
* patients with systemic diseases,
* pregnant women,
* patients who had received MPS treatment within the previous year

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
change from baseline in pain on the 10 point visual analogue scale (VAS) at week 3 | baseline and week 3
  Patients were asked to rate the intensity of their pain on a scale from 0 to 10. They were told that a score of 0 meant no pain, a score of 10 meant severe pain and a score of 5 meant moderate pain
change from baseline in oxygen concentration in the massater muscle at week 3 | baseline and week 3
  oxygen concentration in the massater muscle was measured by functional near-infrared spectroscopy- fNIRS (ARGES cerebro, Hemosoft Inc., Ankara, Turkey) before and after treatment for each patient.
change from baseline in bite force values at week 3 | baseline and week 3
  bite force values were recorded by Flexiforce sensors before and after treatment for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: İREM KARAGÖZOĞLU, Principal Investigator — GAZİANTEP ÜNİVERSİTESİ DİŞ HEKİMLİĞİ FAKÜLTESİ
Locations (1):
- İrem Karagözoğlu, Şehitkamil, Gazi̇antep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karagozoglu I, Demirkol N, Parlar Oz O, Yilmaz S, Ozcan M. New generation low level laser effect on masseter muscle oxygenation, bite force and algometric changes in myofacial pain syndrome: a randomised, placebo-controlled clinical trial. Lasers Med Sci. 2025 Jan 27;40(1):48. doi: 10.1007/s10103-024-04272-z. PMID 39869221